CLINICAL TRIAL: NCT02488733
Title: Laparoscopic Sleeve Gastrectomy Versus Conventional Medical Therapy in Patients With Newly Diagnosed Type 2 Diabetes and Body Mass Index 30-42 Kg/m2: a Randomized Clinical Trial
Brief Title: Early Sleeve Gastrectomy In New Onset Diabetic Obese Patients
Acronym: ESINODOP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Santa Maria, Terni, Italy (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Stefano Trastulli, Azienda Ospedaliera Santa Maria, Terni, Italy, Azienda Ospedaliera Santa Maria, Terni, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESINODOP
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; obesity; laparoscopic sleeve gastrectomy; bariatric surgery; metabolic surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Sleeve Gastrectomy (LSG) (Experimental): In addition to conventional medical therapy, patients assigned to surgical treatment will undergo LSG, to be performed in accordance with current international guidelines.
  Interventions: Procedure: LSG; Drug: CMT
- Conventional medical therapy (CMT) (Other): CMT consists in the use of the best treatment strategies, involving pharmacological and dietary therapies, lifestyle and physical activity, with the aim of both glycemic control and weight loss.
  Interventions: Drug: CMT

INTERVENTIONS:
Procedure: LSG — In addition to all previously described aspects of conventional medical therapy, patients assigned to surgical treatment will undergo LSG, to be performed in accordance with current international guidelines
  Arms: Laparoscopic Sleeve Gastrectomy (LSG)
Drug: CMT — CMT consists in the use of the best treatment strategies, involving pharmacological and dietary therapies, lifestyle and physical activity, with the aim of both glycemic control and weight loss, administered on the basis of the current guidelines of the American Diabetes Association (ADA)[50] and determined on an individual basis [52].The administration of such pharmacological and non-pharmacological therapies will be adjusted in accordance with the algorithms of the ADA .

SUMMARY:
Bariatric surgery is efficient in both inducing adequate weight loss and the control of glycemia in obese patients affected by Type 2 Diabetes Mellitus (T2DM).

Despite growing evidence suggesting that early performance of bariatric surgery on obese patients with T2DM offers the best opportunity to reach and maintain a remission of diabetes, no randomized clinical trials (RCT) have evaluated its efficiency in patients with new T2DM diagnosis.

The aim of this RCT is to compare bariatric surgery, and in particular Laparoscopic Sleeve Gastrectomy (LSG), with conventional medical therapy (CMT) in patients with new T2DM diagnosis that are obese (Body Mass Index, BMI of between 30 and 42 Kg/m2), to be recruited at two Italian diabetology centres (Terni and Rome).

The main objective of the present RCT is to investigate the efficacy of LSG as compared with CMT in inducing and maintaining both a resolution of T2DM (defined as HbA1c levels ≤6.0%, without active pharmacologic therapy or ongoing procedures) and the remission of T2DM through the evaluation of the criteria provided by the American Diabetes Association (ADA) at maximum follow-up of 6 years. The effects of the two treatments in terms of weight loss and the quality of life of the patient will also be taken into consideration.

Any positive results of this study will include preventing microvascular and macrovascular complications connected with diabetes, without the necessity to take medication, and at the same time the loss of excess body weight and improved quality of life (QOL).

DETAILED DESCRIPTION:
Recent evidence suggests that, in obese patients with type 2 diabetes mellitus of long duration, and / or poorly controlled with conventional therapy, bariatric surgery promises diabetes remission rates significantly higher than those attainable with traditional treatment, irrespective of initial BMI and the loss of body weight of the patients.

This has ensured the growing conviction in the international scientific community that bariatric surgery should not be considered as an alternative to conventional obesity and diabetes therapies only after the failure of traditional treatments, but should be performed with the intent to prevent complications associated with these diseases, and therefore at their onset [23]. Furthermore, the use of BMI as the main parameter to guide the indication of bariatric surgery is increasingly being called into question with regard to the presence of comorbidities such as diabetes, as it is the distribution of obesity, together with the presence of comorbidities such as diabetes, rather than the degree of obesity that predicts the onset of related complications.

Bariatric surgery is currently regarded as a "last resort" for both the treatment of obesity and its associated comorbidities, such as diabetes, particularly in patients with a BMI ≤ 35. Despite this, it is now apparent that initial BMI and body weight loss resulting from bariatric surgery have no connection with the metabolic effects of the procedure, such as on the treatment of diabetes. In fact, according to the current national and international guidelines (which are based on a consensus dated 1991[6]), bariatric surgery may be considered in diabetic patients, with a BMI between 30 and 39.9 Kg/m2, only after the recorded failure of conventional medical therapies for obesity and diabetes.

This wait-and-see policy is due to the fact that bariatric surgery is a surgical procedure that is associated, depending on the procedure, with a certain rate of short and long term potential adverse events, and while in the short-medium term it has been shown to achieve significantly higher rates of remission from diabetes, when compared to medical therapy, there remain uncertainties about the durability of remission of diabetes and weight control after long follow-up periods. Essentially, therefore, the risk-benefit ratio has not allowed for the use of bariatric surgery as a first-line therapy for the treatment of type 2 diabetes in obese patients, and in particular in class 1 and 2 obesity. It can be hypothesized, however, that the performance of LSG at diagnosis of diabetes in obese patients can dramatically improve both the resolution/remission rate and the duration of resolution/remission from diabetes, and thus improve the protection against the development of vascular complications.

In fact, growing evidence suggests that the period of time between the diagnosis of diabetes and bariatric surgery is a determining factor in the achievement and duration of diabetes remission. It has also been observed that bariatric surgery is more effective than medical therapy in preventing diabetes in obese patients.

In the opinion of the authors, the early performance of LSG, also at the diagnosis of diabetes, could be crucial. This is hypothesized also on the basis of the well-known phenomenon of "glycemic legacy", according to which the greater the time elapsed between diabetes diagnosis and the achievement, with any form of therapy, of glycemic control targets, the lower the benefit in terms of protection from the development of vascular complications associated with diabetes [34]. It follows that blood glucose control in patients with newly diagnosed diabetes should be achieved through the implementation of appropriate treatments, including bariatric surgery, as quickly as possible after diagnosis. In this sense, bariatric surgery (and in particular, LSG) has been proven capable of promoting glycemic control in the short to medium term, in terms of the substantial and rapid reduction of glycated haemoglobin, (even 3 months after surgery), compared to conventional medical therapy in patients with longstanding diabetes (about 9 years on average). In the RCT conducted by Schauer et al., 3 months after sleeve gastrectomy, average HbA1c levels were reduced from an initial average value of 9.5% to 7%, while in the medical-therapy group they were reduced from an initial value of 8.9% to 7.7%,therefore significantly less effective than LSG. Thus irrespective of the rate of achievement and duration of eventual remission of diabetes (that in any case is already at present considerably higher than medical therapy in patients with longstanding and poorly controlled diabetes), patients undergoing sleeve gastrectomy (and bariatric surgery in general) could benefit from the procedure being performed on diagnosis of diabetes, and therefore as soon as possible, thanks to the ability to reach the HbA1c target level for glycemic control more easily and quickly than with medical therapy. This would have a proven protective effect on long-term vascular complications, irrespective of the duration of the glycemic control and the achievement of any remission on the basis of the concept of "glycemic legacy" and "metabolic memory" , through the analysis of the results of the largest and most prestigious international randomized clinical trials on the treatment of diabetes (UKPDS, DCCT/EDIC, ACCORD and VATD trials).

The phenomenon of metabolic memory refers to the fact that the UKPDS and DCCT / EDIC studies have demonstrated that even a transitory period of aggressive glycemic control, such as that attainable after bariatric surgery, is capable of inducing a beneficial "metabolic memory", with the effect of reducing microvascular complications over time, regardless of subsequent maintenance of glycemic control [32].

Then the rationale for the use of bariatric surgery at diagnosis of type 2 diabetes mellitus is based not only on the hypothesis of the attainment of early and sustained glycemic control in obese patients, but also on a variety of scientific evidence that suggests that the precocity of its performance is a positive predictor of remission and of the long-term maintenance of diabetes remission.

As previously mentioned, the superiority of bariatric surgery to conventional medical therapy in obese patients (even with BMI less than 30) with diabetes of long duration, and / or poorly controlled with conventional therapy, in terms of attaining glycemic control, has clearly been demonstrated , even if for medium-short follow-up periods [1]. When applied in obese patients with new onset diabetes it might therefore subvert the risk-benefit ratio that now prevents its use as a first-line therapy, thanks to an increase in the rate of remission of diabetes and its endurance, as well as a reduction of the long-term vascular complications of diabetes.

In conclusion, a recent American Society of Metabolic and Bariatric Surgery (ASMBS) position statement noted that that class 1 obesity requires effective treatment, as it represents a significant health problem, and that treatment should involve the use of bariatric surgery. Indeed, recent randomized studies have demonstrated both the effectiveness, in terms of weight loss and control of comorbidity, and the safety of some bariatric surgical procedures, including sleeve gastrectomy, in this specific group of patients (Class 1 Obesity).

These observations suggest that T2DM could be treated with bariatric surgery as early as possible, also at the time of diagnosis.

It can be hypothesized that performing LSG at T2DM diagnosis can offer the maximum benefits in terms of both the attainment and duration of T2DM resolution/remission, with the potential to thus prevent micro and macrovascular complications without the need to take medication. Other positive aspects include the possibility to achieve appropriate weight loss and a related improvement in the quality of life. In this randomized trial LSG will be compared with conventional medical therapy in the treatment of T2DM at onset in obese patients with a BMI of between 30 and 42 Kg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. No contraindication for laparoscopic surgery or general anaesthesia.
2. Age ≥20 and ≤65 years.
3. BMI of between 30 and 42 kg/m2.
4. Documented new diagnosis of Type 2 Diabetes Mellitus obtained according to the following American Diabetes Association parameters: fasting blood glucose ≥ 126 mg/dl (7.0 mmol/l) and/or HbA1c ≥ 6.5% and no more than 8 months from enrollment in the study.

Exclusion Criteria:

1. Previous bariatric surgery or major abdominal surgery.
2. Patients with T2DM diagnosis treated with insulin.
3. Evidence of complications connected to diabetes at any stage (diabetic retinopathy, diabetic nephropathy/microalbuminuria, cardiovascular disease or neuropathy).
4. Cardiovascular diseases such as ischemia / coronary artery disease, arrhythmia, peripheral vascular diseases, congestive heart failure, history of heart attacks.
5. Kidney diseases including nephro-vascular hypertension, stenosis of the renal artery or chronic renal insufficiency.
6. Pregnancy
7. Diagnosis of psychiatric illness (including dementia, severe depression, history of suicide attempts) or abuse of alcohol or drugs in the previous 5 years.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients achieving diabetes resolution | Assessed up to 1 year after randomization
  HbA1c levels ≤6.0%, without active pharmacologic therapy or ongoing procedures

SECONDARY OUTCOMES:
Rate of patients achieving diabetes resolution | assessed at 2, 3, 4, 5 and 6 years after randomization
  diabetes resolution
Rate of patients achieving diabetes complete remission (American Diabetes Association criteria) | assessed at 2, 3, 4, 5, and 6 years after randomization
  diabetes complete remission
Rate of patients achieving HbA1c levels ≤6.5%, | assessed at 1, 2, 3, 4, 5,and 6 years after randomization
  achieving HbA1c levels ≤6.5%,
Rate of patients achieving HbA1c levels ≤6.5%, | assessed up at 1, 2, 3, 4, 5,and 6 years after randomization
  achieving HbA1c levels ≤6.5%,
Rate of patients achieving prolonged remission (American Diabetes Association criteria) | Assessed up at 6 years after randomization
  achieving prolonged remission
Time to achievement (in days) of complete remission | Assessed up at 2 years after randomization
  complete remission
Time to achievement (in days) of prolonged remission | Assessed up at 6 years after randomization
  prolonged remission
Total duration of the period with diabetes resolution | Assessed at 3 and 6 years
  diabetes resolution
Total duration of the period in complete remission | Assessed at 3 and 6 years
  complete remission
Total duration of the time period with HbA1c ≤ 6.0% irrespective of any active pharmacologic therapy or ongoing procedures | Assessed at 3 and 6 years
  Total duration of the time period with HbA1c ≤ 6.0% irrespective of any active
Total duration of the period with HbA1c levels ≤6.5%, without active pharmacologic therapy or ongoing procedures | Assessed at 3 and 6 years
  Total duration of the period with HbA1c levels ≤6.5%, without active pharmacologic
Total duration of the period with HbA1c levels ≤6.5% irrespective of any active pharmacologic therapy or ongoing procedures | Assessed at 3 and 6 years
  Total duration of the period with HbA1c levels ≤6.5% irrespective of any active
Average value and changes from baseline, during the follow-up period, until the predefined time end-points of anthropometric, blood, urinary and QoL parameters. | Assessed up at 6 years after randomization
  Average value and changes from baseline, during the follow-up period, until the
Rate of patients with effective weight loss (defined as % Excess Weight Loss > 50%) | Assessed at 2 ,4, 6 years after randomization
  Rate of patients with effective weight loss (defined as % Excess Weight Loss > 50%)
Rate of patients with hypertension and / or requiring antihypertensive therapy | Assessed at 2,4, 6 years after randomization
  Rate of patients with hypertension and / or requiring antihypertensive therapy
Rate of patients with dyslipidemia and / or that require drug therapy for dyslipidemia | Assessed at 2,4 6 years after randomization
  Rate of patients with dyslipidemia and / or that require drug therapy for dyslipidemia
Complications related to diabetes, or its pharmacological treatment, as well as those resulting from bariatric surgery. | Assessed at 2,4 6 years after randomization
  Complications related to diabetes, or its pharmacological treatment, as well as those
Renal (onset of nephropathy or microalbuminuria), cardiovascular (defined as the occurrence of myocardial infarction, congestive heart failure or stroke), and ocular damage (development of diabetic retinopathy), and diabetes-related peripheral neuropathy | Assessed at 2,4, 6 years after randomization
  Renal (onset of nephropathy or microalbuminuria), cardiovascular (defined as the occurrence of myocardial infarction, congestive heart failure or stroke), and ocular damage (development of diabetic retinopathy), and diabetes-related peripheral neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Trastulli, MD, Principal Investigator — Azienda Ospedaliera Santa Maria di Terni
Locations (2):
- Italy (2):
  - Ospedale Sandro Pertini, Rome
  - Azienda Ospedaliera Santa Maria, Terni

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official study website — https://esinodop.logix-software.it